CLINICAL TRIAL: NCT05740800
Title: Patient Care Needs and the Decision-Making Experience of Patients With Cancer and Family Caregivers Regarding Immunotherapy: A Qualitative and Quantitative Mixed Methods Study
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201812191RINB
Record Dates: First submitted 2022-01-13; First posted 2023-02-23 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2023-02

CONDITIONS: Supportive Care Needs; Immunotherapy
Keywords: cancer; caregiver; immune therapy; treatment decision making; care need
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Immunotherapy is currently a crucial cancer treatment option. Despite the development of new cancer treatment, patients and their family caregivers still experience complex psychological feelings and challenges about the effectiveness of immunotherapy, financial burden, and treatment related side effects which reflect the problems related to decision-making and the supportive care needs.

ELIGIBILITY:
Patient

Inclusion Criteria:

1. 20 years old and above.
2. Patients diagnosed with cancer by a physician.
3. The patient has a known condition and has received immunotherapy.
4. Those who have received at least 1 time immunotherapy, including: receiving a single drug or immunotherapy combined with other treatment.

Exclusion Criteria:

1. Patients with mental illness.
2. Confused and unable to communicate verbally or in writing to complete the research interviews.
3. Those who are reluctant to accept interviews and participate in research surveys.

Family caregivers

Inclusion Criteria:

1. 20 years old and above.
2. Live with the patient and spend the most time caring for the patient.
3. The primary family caregiver is identified by the patient.

Exclusion Criteria:

1. Caregivers with mental illness.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cancer patients and their family caregivers with immunotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Supportive Care Needs Survey | 1 time points: From date of approaching patient until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Patients' and family caregivers' supportive care needs will be measured by Supportive Care Needs Survey(SCNS) .It is a 5-Point Likert Scale,higher scores mean more care needs.

SECONDARY OUTCOMES:
Physical and Psychological Symptoms Scale | 1 time points: From date of approaching patient until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Patients' and family caregivers' physical and psychological symptoms will be measured by Physical and Psychological Symptom Scale.It use Numerical Rating Scale(VRS)0-10.It is a 11 Point Likert Scale(e. g. 0 is no pain; 10 is unbearable pain) .
CollaboRATE scale and SURE scale | 1 time points: From date of approaching patient until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Patients' and family caregivers' decision making process and conflict will be measured by CollaboRATE scale and SURE scale. CollaboRATE scale is a 10-Point Likert Scale (0-9), higher the score, the more effort you pay on this issues. SURE scale which base on Decisional Conflict Scale are 4 items,The question you agree that you can answer "YES" and got 1 point,if you not fit the description you have to answer "NO" and got 0 points,The lower the total score, the greater the decision conflict.
Comprehensive Score for Financial Toxicity-Functional Assessment of Chronic Illness Therapy (COST-FACIT) | 1 time points: From date of approaching patient until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Patients' financial toxicity will be measured by COST-FACIT. It is a 5-Point Likert Scale (0-4),The higher the score for each question, the more often the problem occurs.
Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 1 time points: From date of approaching patient until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Patients' immunotherapy side effects will be measured by CTCAE.The severity is divided into 5 grades, the higher the grade, the higher the severity.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Taipei, Taiwan